CLINICAL TRIAL: NCT03326505
Title: The Effect of Stem Cell Therapy and Comprehensive Physical Therapy in Motor and Non-Motor Symptoms in Patients With Multiple Sclerosis: A Comparative Study.
Brief Title: Allogenic Mesenchymal Stem Cells And Physical Therapy for MS Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Fatima Jamali, Head of Neuroscience Research, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALLOMSUJCTC
Record Dates: First submitted 2017-05-09; First posted 2017-10-31 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Umbilical Cord Mesenchymal Stem Cells; Multiple Sclerosis; Neuroimmunology; Autoimmune disease; Physical therapy
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Injection of Umbilical cord derived UC- MSCs (Active Comparator): Allogenic Umbilical Cord derived stem cells injected intrathecally to enrolled MS patients
  Interventions: Biological: Umbilical cord derived Mesenchymal Stem Cells
- injection of UC- MSCs and SPT (Active Comparator): Allogenic Umbilical Cord derived stem cells injected intrathecally to enrolled MS patients along with a supervised physical therapy program
  Interventions: Biological: Umbilical cord derived Mesenchymal Stem Cells; Other: Supervised physical therapy
- Supervised Physical Therapy (SPT) (Active Comparator): Supervised physical therapy program without stem cells
  Interventions: Other: Supervised physical therapy

INTERVENTIONS:
Biological: Umbilical cord derived Mesenchymal Stem Cells — Allogenic umbilical cord derived stem cells which are to be injected intrathecally as a treatment option for consenting MS patients
  Other Names: UC-MSCs
  Arms: Injection of Umbilical cord derived UC- MSCs; injection of UC- MSCs and SPT
Other: Supervised physical therapy — A combined physical therapy program of Balance, strengthening and endurance exercises
  Other Names: SPT
  Arms: Supervised Physical Therapy (SPT); injection of UC- MSCs and SPT

SUMMARY:
This study aims at expanding Umbilical Cord derived Mesenchymal Stem Cells (MSCs) to a clinical scale according to Good Laboratory Practice and study its efficacy when compared to a Supervised Physical Therapy Program alone.

DETAILED DESCRIPTION:
Umbilical cord derived MSCs bank will be generated and all patients given the same cells from the same biological sample.

Thorough clinical, cognitive and motor analysis will be performed at baseline and compared to outcomes at 3 different time points of all enrolled patients.

The study will consist of three arms: 1- Stem cells treatment 2- Stem cells and supervised physical therapy 3- Supervised physical therapy

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of definite MS according to the revised McDonald Criteria.
* Expanded Disability Status Scale (EDSS) ≤ 7
* Failure of standard medical therapy
* Disease duration of at least three years prior to enrollment.

Exclusion Criteria:

* Pregnant and lactating women
* Previous treatment with immunosuppressive agents in the last 12 months prior to enrollment
* Recent MS relapse in the month prior to enrollment
* Treatment with oral or parenteral steroids for any cause in the month prior to enrollment
* Significant systemic medical disorders including cardiac, renal, hepatic, hematologic, immunologic or endocrine disorders
* Previous treatment with interferons or glatiramer acetate in the 3 months prior to enrollment
* Any contra-indication for magnetic resonance imaging (MRI) or gadolinium contrast.
* Positive serology for HIV, Hepatitis B or Hepatitis C
* Any history of malignancy or exposure to radiation at any time prior to enrollment
* Any contra-indication to lumbar puncture
* Severe cognitive impairment that would interfere with the patient's ability to understand and sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Isolation and Expansion of Mesenchymal Stem Cells | 3-6 months
  To isolate stem cells from UC: first, the cord will be cut into small pieces around (4-5cm) and washed with phosphate buffered saline, then the umbilical vein and the two arteries will be removed.These pieces will be placed in culture plate and cultured in UC-MSCs medium consist of; alpha modification of Minimum Essential Medium (α-MEM) supplemented with 10% fetal bovine serum, 1% glutamine, 1% penicillin/streptomycin and 1 μg/mL amphotericin B.After incubation period the undigested tissue will be discarded and nucleated cells will be pelleted by centrifugation at 450xg for 10 minutes. Cell pellet will be re-suspended in UC-MSCs culture medium, cultured in tissue culture flasks and placed in CO2 incubator at 37°C, 5% CO2. Cells will be expanded in multilayer cell factory tissue culture flasks to reach an estimated 108 UC-MSCs that will be frozen in bags of 106 cells for subsequent thawing and administration.

SECONDARY OUTCOMES:
Safety and Efficacy Assessment Pre and Post Treatment | 3-12 months
  Outcome measures will be assessed at 3 months pre-treatment, baseline (prior injections), 3 months, 6 months, and 12 months.
  Informed consent will be obtained in writing from each subject prior to participation in the study. If the subject is unable to give consent or he/she scores less than 24 on the Mini Mental Status Examination (MMSE), they will be excluded from the study. The research personnel involved in the study will carefully explain the consent form to the subject. The subject will then be given ample opportunity to ask questions prior agreeing to participate. If the need arises the research personnel will be available to answer questions and address any concerns.
Motor Functions Assessments | 3-12 months
  A number of motor function tests will be performed with every follow up visit for all 30 patients.
Measuring Non-motor outcomes to assess treatment efficacy. | 3-6 months
  Clinical Tests ,all patients will be evaluated clinically using qualitative and quantitative tests.
Biological Assessments | 3-12 months
  Blood samples will be collected pre and post treatment for immediate or ulterior analysis. Results will be compared between individuals and then between the two groups that received one or two doses of UC-MSCs.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center
Locations (2):
- Jordan (2):
  - Cell Therapy Center, University of Jordan, Amman
  - Cell Therapy Center, Amman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alghwiri AA, Jamali F, Aldughmi M, Khalil H, Al-Sharman A, Alhattab D, Al-Radaideh A, Awidi A. The effect of stem cell therapy and comprehensive physical therapy in motor and non-motor symptoms in patients with multiple sclerosis: A comparative study. Medicine (Baltimore). 2020 Aug 21;99(34):e21646. doi: 10.1097/MD.0000000000021646. PMID 32846775